CLINICAL TRIAL: NCT02127164
Title: Prospective Evaluation of Wound Management Using Vacuum Assisted Instillation Therapy in Emergent Contaminated Abdominal Surgeries
Brief Title: Vacuum Assisted Therapy in Emergent Contaminated Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Andrew Tang, Assistant Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAKCI2014
Record Dates: First submitted 2014-04-04; First posted 2014-04-30 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Injury; Complicated Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "Veraflo" device, Dakin's solution (Experimental)
  Interventions: Device: "Veraflo" device, Dakin's solution

INTERVENTIONS:
Device: "Veraflo" device, Dakin's solution — Veraflo device will be installed on the wound to create negative pressure after surgery. Dakin's solution will be instilled through this device into the wound at the regular intervals.

SUMMARY:
Emergent abdominal surgeries have very high rate of wound contamination due to exposure to bacteria from GI tract. There are several different approaches to wound management in these patients including wet-to-dry dressing or application vacuum assisted device on the wound. The investigators propose using the vacuum assisted device with Dakin's solution on patients undergoing emergency surgery for hollow viscus perforation installed immediately at the end of operation and remained there for the first 3 postoperative days, followed by delayed primary closure on postoperative day 4. The investigators believe this technique can achieve earlier wound closure, decrease patient discomfort, improve cost savings, and potentially standardize and revolutionize the investigators management of heavily contaminated wounds.

ELIGIBILITY:
Inclusion Criteria:

* Emergent surgery involving hollow viscus perforation or necrotic bowel
* Admitted to the University of Arizona Medical Center, Tucson, AZ

Exclusion Criteria:

* Prisoners
* Pregnancy
* Patients with allergy to Dakin's (sodium hypochlorite) solution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Tang, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Veraflo" Device, Dakin's Solution
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | "Veraflo" Device, Dakin's Solution
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.8)
Smokers [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of Surgical Site Infection
Description: Surgical site infection is defined as the presence of localized inflammatory signs such as hyperthermia, erythema, tenderness, or purulent discharge that results in positive cultures, along with positive wound cultures. Surgical site can also be regarded as infected based on the individual discretion of the treating physician. Surgical sites with >10^5 colonization in swab will be considered contaminated.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | "Veraflo" Device, Dakin's Solution
Number analyzed (Participants) | 18
Participants | 5

2. Secondary Outcome: Wong-Baker Faces Pain Rating Scale
Description: The Wong-Baker Faces Pain Rating scale is used to grade pain related to the presence/manipulation of the device. The Wong-Baker scale range is from 0 (No Hurt) to 10 (Hurts Worst) with numbers increasing by 2 (0, 2, 4, 6, 8, 10) and associated face images showing increased pain and sadness. Higher scores indicate increased pain, a worse outcome.
Time Frame: 1 week
Measure: Mean (Full Range); unit: pain score
Arm/Group | "Veraflo" Device, Dakin's Solution
Number analyzed (Participants) | 18
pain score | 6 [4 to 6]

ADVERSE EVENTS:
Time Frame: Through hospital discharge (approx. 2 weeks)
Arm/Group | "Veraflo" Device, Dakin's Solution
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Limited sample size as a result of difficulty in consenting subjects prior to trauma surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT02127164/Prot_SAP_000.pdf